CLINICAL TRIAL: NCT04249505
Title: The Refractive Accuracy of Photoscreeners "2WIN" and "PlusoptiX" and the "Retinomax" Auto Refractor
Brief Title: Refractive Accuracy of "2WIN" and Portable Autorefractors
Status: Completed | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: ABCD RefAcc
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2020-07

CONDITIONS: Refractive Error - Myopia Axial; Astigmatism; Accomodation; Visual Impairment; Hyperopia of Both Eyes
Keywords: photoscreening; photo refraction; auto refraction; spectacle dispensing
MeSH Terms: conditions — Astigmatism; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: "2WIN" Photoscreener — non-cycloplegia refraction by Adaptica "2WIN"
Device: "Plusoptix A12" — non-cycloplegic refraction by "Plusoptix A12" photoscreener
Device: "Retinomax" — non-cycloplegic refraction by "Retinomax K+" auto refractor

SUMMARY:
Youth and some adults have photoscreening refractions and hand-held auto refraction before cycloplegia refraction during new and follow up eye examinations. Vector math is applied to each refraction to determine how closely the hand-held "dry" devices match actual refraction.

DETAILED DESCRIPTION:
A closeness-of-fit algorithm utilizing vector transformations of astigmatism is designed and applied to 50-years of clinical international refractive experience.

As a part of new and follow up comprehensive eye examinations, patients and parents consented to confirm the cycloplegic refraction to other portable refractive tools.

The ability of photoscreeners "2WIN" ("Adaptica," Padova italy), "PlusoptiX A12" (Nuremberg, Germany) and "Retinomax" (Righton, Tokyo, Japan) to match actual refraction is assessed utilizing the new algorithm.

This algorithm could then be applied to batches of donated spectacles distend by charitable organizations worldwide if portable auto refracting devices are employed.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing new or follow examination at pediatric eye and adult strabismus clinic Willing to undergo screening refractive device developmental delays included

Exclusion Criteria:

* Intraocular lens in place

Ages: 6 Months to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: children and adults attending pediatric ophthalmology and adult strabismus clinic
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Refractive Accuracy | 1 day
  spherical equivalent
Refractive Accuracy | 1 day
  Vector transform J0 and J45 astigmatism
Refractive Accuracy | 1 day
  Spectacle comparison score (Percent similarity combined sphere-cylinder)

SECONDARY OUTCOMES:
Impact of age | 1 day
  Spectacle similarity score striated by age relative to patient's ability to accommodate

CONTACTS AND LOCATIONS:
Overall Officials: Bob Arnold, MD, Principal Investigator — Coordinator Alaska Blind Child Discovery
Locations (1):
- Alaska Children's EYE & Strabismus, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified database shared on www.ABCD-Vision.org Website.
Supporting Information: Analytic Code
Time Frame: after study completed
Access Criteria: open
URL: http://www.abcd-vision.org/references/index.html

REFERENCES:
- [Background] Arnold SL, Arnold AW, Sprano JH, Arnold RW. Performance of the 2WIN Photoscreener With "CR" Strabismus Estimation in High-Risk Patients. Am J Ophthalmol. 2019 Nov;207:195-203. doi: 10.1016/j.ajo.2019.04.016. Epub 2019 May 9. PMID 31077668